CLINICAL TRIAL: NCT03627065
Title: An Open-Label Phase 2 Study of INCB050465 in Participants With Primary Sjögren's Syndrome
Brief Title: A Study of INCB050465 in Primary Sjögren's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 50465-207; Parsaclisib (Other: Incyte Corporation)
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Results first posted 2021-03-24 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Primary Sjögren's Syndrome
Keywords: Primary Sjögren's syndrome; PI3Kδ inhibitor
MeSH Terms: interventions — parsaclisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Parsaclisib (Experimental)
  Interventions: Drug: Parsaclisib

INTERVENTIONS:
Drug: Parsaclisib — Parsaclisib administered orally once daily at the protocol-defined dose.
  Other Names: INCB050465

SUMMARY:
The purpose of this study is to assess the impact of parsaclisib on the signs and symptoms of Sjögren's syndrome (SS).

ELIGIBILITY:
Inclusion Criteria:

* Primary SS diagnosed according to the revised American-European Consensus Group (AECG) criteria.
* Minimum score of 2 on the SGUS score for parotid and submandibular glands.
* EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) score ≥ 5.
* Positive serum titers of anti-SS-A and/or anti-SS-B antibodies.
* Symptomatic oral dryness score of at least 5 on patient questionnaire.
* Willingness to avoid pregnancy or fathering children based on protocol-defined criteria.

Exclusion Criteria:

* Diagnosis of secondary SS according to the revised AECG criteria (eg, the presence of a previously diagnosed or a present diagnosis of rheumatoid arthritis, systemic lupus erythematosus, systemic sclerosis, mixed connective tissue disease, polymyositis, dermatomyositis, immunoglobulin G4-related disorder, sarcoidosis, or any other defined autoimmune rheumatologic disorder).
* Concurrent conditions and history of other diseases per protocol-defined criteria.
* Positive test results for tuberculosis (TB) from the QuantiFERON-TB Gold test or T-spot.TB test.
* Positive serology test results for HIV antibody, hepatitis B surface antigen, hepatitis B surface antigen antibody, HBV core antibody, or HCV (HCV antibody with positive HCV-RNA).
* Severely impaired liver function (Child-Pugh Class C).
* Prior or ongoing therapy with protocol-defined drugs.
* Receipt of any live vaccine in the 30 days before screening.
* No major surgery within 30 days before screening. Inadequate recovery from toxicity and/or complications from a major surgery before starting therapy.
* Current alcohol or drug use that, in the opinion of the investigator, will interfere with the participant's ability to comply with the dose regimen and study evaluations.
* Laboratory values at screening outside the protocol-defined ranges.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-12-07 (Actual); Study Completion 2020-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Butler, MD, Study Director — Incyte Corporation
Locations (4):
- United States (4):
  - Advanced Pharma CR, Miami, Florida
  - North Georgia Rheumatology Group, Lawrenceville, Georgia
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Ramesh C. Gupta, MD, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 12 participants were planned. Ten participants were enrolled and analyzed for efficacy and safety.
Pre-assignment Details: Ten participants were enrolled and treated. Seven participants completed treatment. Three participants discontinued treatment and withdrew from the study.
Groups:
- Parsaclisib: parsaclisib was administered orally once a day.
Period: Overall Study
Arm/Group | Parsaclisib
Started | 10
Completed | 7
Not Completed | 3
Not completed — Study Terminated by sponsor | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Parsaclisib: parsaclisib was administered orally once a day for up to 12 weeks.
Arm/Group | Parsaclisib
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.1 (13.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 4
  Black/African-American | 6

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With a 1 Point or Greater Change on the Salivary Gland Ultrasound (SGUS) Score for Parotid and Submandibular Glands
Description: The SGUS is a combination of the scores of the 4 salivary glands (2 parotid and 2 submandibular) each gland is scored on a 5-point scale (0 to 4; 4 being more severe), with the maximum total score being 16.
Time Frame: Week 4 and Week 12
Population: Full analysis set included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Parsaclisib
Number analyzed (Participants) | 10
Participants
  Week 4: number analyzed (Participants) | 8
  Week 4 | 0
  Week 12: number analyzed (Participants) | 7
  Week 12 | 0

2. Secondary Outcome: Change From Baseline in Salivary CXCL13 Levels
Description: To assess the impact of parsaclisib on salivary CXCL13.
Time Frame: Baseline, Week 4 and Week 12
Population: Full analysis set included all participants enrolled in the study who received at least 1 dose of study drug, and detectable levels of CXCL13.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Parsaclisib
Number analyzed (Participants) | 2
L/h
  Week 4 | 0.96 (0.1)
  Week 12 | 1.98 (1.4)

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug.
Time Frame: Up to 21 weeks
Population: The full analysis set included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Parsaclisib
Number analyzed (Participants) | 10
Participants | 4

4. Secondary Outcome: Change in Whole Salivary Flow
Description: Defined as change in stimulated and unstimulated whole salivary flow from baseline
Time Frame: Baseline, Weeks 4, 8, and 12
Population: The full analysis set included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: g/min
Arm/Group | Parsaclisib
Number analyzed (Participants) | 10
g/min
  Mean change in stimulated salivary flow Week 4: number analyzed (Participants) | 9
  Mean change in stimulated salivary flow Week 4 | 0.07 (0.152)
  Mean change in stimulated salivary flow Week 8: number analyzed (Participants) | 6
  Mean change in stimulated salivary flow Week 8 | -0.05 (0.129)
  Mean change in stimulated salivary flow Week 12: number analyzed (Participants) | 7
  Mean change in stimulated salivary flow Week 12 | -0.05 (0.144)
  Mean change in unstimulated salivary flow Week 4: number analyzed (Participants) | 9
  Mean change in unstimulated salivary flow Week 4 | 0.03 (0.046)
  Mean change in unstimulated salivary flow Week 8: number analyzed (Participants) | 6
  Mean change in unstimulated salivary flow Week 8 | 0.07 (0.109)
  Mean change in unstimulated salivary flow Week 12: number analyzed (Participants) | 7
  Mean change in unstimulated salivary flow Week 12 | 0.04 (0.082)

5. Secondary Outcome: Change in EULAR Sjögren's Syndrome Disease Activity Index
Description: Defined as change in ESSDAI. The ESSDAI is a physician-assessed disease activity index for primary Sjögren's syndrome developed by the EULAR consortium. It consists of 44 items in 12 organ-specific 'domains' contributing to disease activity (constitutional, lymphadenopathy, articular, muscular, cutaneous, glandular, pulmonary, renal, peripheral nervous system, central nervous system, hematological, biological). Each domain is assessed for activity level (i.e., no, low, moderate, high) and assigned a numerical score based on pre-determined weighting of each individual domain. An overall score is then calculated as the sum of all individual weighted domain scores. Overall score is calculated as sum of all individual weighted domain scores (ranges from 0 (best) to 123 (worst activity).
Time Frame: Week 12
Population: Full analysis set included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Parsaclisib
Number analyzed (Participants) | 10
Index
  Mean Change at Week 4: number analyzed (Participants) | 9
  Mean Change at Week 4 | -0.3 (2.92)
  Mean Change at Week 8: number analyzed (Participants) | 7
  Mean Change at Week 8 | -2.0 (4.12)
  Mean Change at Week 12: number analyzed (Participants) | 7
  Mean Change at Week 12 | -5.3 (4.15)

6. Secondary Outcome: Change in EULAR Sjögren's Syndrome Patient Reported Index
Description: Defined as Change in ESSPRI. EULAR Sjogren's Syndrome Patient-Reported Index (ESSPRI) Score is defined as the change in score between baseline (Week -1) and Week 12. The ESSPRI is a patient-reported, subjective symptom index for primary Sjögren's syndrome developed by the EULAR consortium. It consists of three questions covering the cardinal symptoms of Sjögren's syndrome: dryness, fatigue and pain (articular and/or muscular). Each domain scored on scale of 0-10 (0 =no symptom at all and 10 = worst symptom imaginable), and an overall score is calculated as the mean of the three individual domains where all domains carry the same weight.
Time Frame: Weeks 4, 8, and 12
Population: Full analysis set included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Parsaclisib
Number analyzed (Participants) | 9
Index
  Mean Change at Week 4 | -1.9 (2.26)
  Mean Change at Week 8: number analyzed (Participants) | 7
  Mean Change at Week 8 | -2.0 (1.93)
  Mean Change at Week 12: number analyzed (Participants) | 7
  Mean Change at Week 12 | -1.8 (1.98)

7. Secondary Outcome: Change in Symptom Scores for Dryness
Description: Defined as change in symptom scores for dryness of eyes, mouth, and vagina. The dryness questionnaire will ask participants to rate the dryness of eyes, mouth, or vagina (female participants only) with 24-hour recall using an 11-point numerical rating system ranging from 0 (no dryness) to 10
Time Frame: Weeks 4, 8, and 12.
Population: Full analysis set included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Parsaclisib
Number analyzed (Participants) | 10
Scores on a scale
  Change in Symptom Score for eye dryness at Week 4: number analyzed (Participants) | 9
  Change in Symptom Score for eye dryness at Week 4 | -2.6 (2.96)
  Change in Symptom Score for eye dryness at Week 8: number analyzed (Participants) | 7
  Change in Symptom Score for eye dryness at Week 8 | -2.4 (2.07)
  Change in Symptom Score for eye dryness at Week 12: number analyzed (Participants) | 7
  Change in Symptom Score for eye dryness at Week 12 | -2.4 (2.64)
  Change in Symptom Score for mouth dryness at Week 4: number analyzed (Participants) | 9
  Change in Symptom Score for mouth dryness at Week 4 | -2.8 (2.64)
  Change in Symptom Score for mouth dryness at Week 8: number analyzed (Participants) | 7
  Change in Symptom Score for mouth dryness at Week 8 | -2.1 (2.41)
  Change in Symptom Score for mouth dryness at Week 12: number analyzed (Participants) | 7
  Change in Symptom Score for mouth dryness at Week 12 | -3.6 (2.99)
  Change in Symptom Score for vaginal dryness at Week 4 | -1.3 (3.20)
  Change in Symptom Score for vaginal dryness at Week 8 | -2.3 (3.50)
  Change in Symptom Score for vaginal dryness at Week 12 | -1.3 (2.94)

8. Secondary Outcome: Patient Global Impression of Change Questionnaire
Description: Defined as proportions of participants in each PGIC category. The PGIC asks a single question regarding how the patient is feeling since beginning new therapy. The questionnaire uses a 7-point scale (from 1 to 7), ranging from "very much improved, 1" to "very much worse, 7
Time Frame: Baseline, Weeks 4, 8, and 12
Population: Full analysis set included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Parsaclisib
Number analyzed (Participants) | 10
Participants
  Baseline: number analyzed (Participants) | 9
  Baseline: Very Much Worse | 0
  Baseline: Worse | 0
  Baseline: Somewhat Worse | 0
  Baseline: No Change | 9
  Baseline: Somewhat Improved | 0
  Baseline: Improved | 0
  Baseline: Very much Improved | 0
  Week 4: number analyzed (Participants) | 9
  Week 4: Very Much Worse | 0
  Week 4: Worse | 0
  Week 4: Somewhat Worse | 0
  Week 4: No Change | 3
  Week 4: Somewhat Improved | 2
  Week 4: Improved | 4
  Week 4: Very much Improved | 0
  Week 8: number analyzed (Participants) | 7
  Week 8: Very Much Worse | 0
  Week 8: Worse | 0
  Week 8: Somewhat Worse | 0
  Week 8: No Change | 2
  Week 8: Somewhat Improved | 2
  Week 8: Improved | 3
  Week 8: Very much Improved | 0
  Week 12: number analyzed (Participants) | 7
  Week 12: Very Much Worse | 0
  Week 12: Worse | 0
  Week 12: Somewhat Worse | 0
  Week 12: No Change | 2
  Week 12: Somewhat Improved | 2
  Week 12: Improved | 3
  Week 12: Very much Improved | 0

9. Secondary Outcome: Change in PROMIS Fatigue Short Form
Description: Defined as change in PROMIS Fatigue short form. The PROMIS fatigue short form includes 7 items with a rating scale of 1 to 5, 1 being no fatigue and 5 being severe fatigue. The recall period is 7 days.
Time Frame: Weeks 4, 8, and 12
Population: Full analysis set included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Parsaclisib
Number analyzed (Participants) | 10
Scores on a scale
  Change in Score at Week 4: number analyzed (Participants) | 9
  Change in Score at Week 4 | -2.6 (4.03)
  Change in Score at Week 8: number analyzed (Participants) | 7
  Change in Score at Week 8 | -1.9 (2.79)
  Change in Score at Week 12: number analyzed (Participants) | 7
  Change in Score at Week 12 | -1.7 (2.87)

10. Secondary Outcome: Female Participants Only : Change in Female Sexual Function Index
Description: Defined as change in FSFI. The FSFI is a brief, self-report measure of female sexual function (female participants only). The questionnaire contains 19 item sexual functioning questionnaire to rate sexual function between 2.0 and 36.0, where 2.0 is low sexual function and 36.0 is high sexual function. Difference in FSFI scores are reported.
Time Frame: Weeks 4, 8, and 12
Population: Full analysis set included all female participants enrolled in the study who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Parsaclisib
Number analyzed (Participants) | 9
Index
  Change in Functional Index at Week 4: number analyzed (Participants) | 8
  Change in Functional Index at Week 4 | 1.8 (3.19)
  Change in Functional Index at Week 8: number analyzed (Participants) | 6
  Change in Functional Index at Week 8 | 2.8 (4.76)
  Change in Functional Index at Week 12: number analyzed (Participants) | 6
  Change in Functional Index at Week 12 | 1.3 (1.83)

11. Secondary Outcome: Change in European Quality of Life 5 Dimensions Questionnaire
Description: Defined as change in EQ-5D. The EQ-5D is a standardized measure of health status. It consists of 5 questions, each with a 5-item rating scale plus a visual analog scale rating from 1 to 100 for overall health status. Higher score represents more severe symptoms.
Time Frame: Weeks 4, 8, and 12
Population: Full analysis set included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Parsaclisib
Number analyzed (Participants) | 10
Scores on a scale
  Change in EQ5D at week 4: number analyzed (Participants) | 9
  Change in EQ5D at week 4 | 7.2 (17.34)
  Change in EQ5D at week 8: number analyzed (Participants) | 7
  Change in EQ5D at week 8 | 0.7 (28.05)
  Change in EQ5D at week 12: number analyzed (Participants) | 7
  Change in EQ5D at week 12 | -6.4 (22.49)

12. Secondary Outcome: Percentage Change in Whole Salivary Flow
Description: Defined as change and percent change in stimulated and unstimulated whole salivary flow from baseline
Time Frame: Baseline, Weeks 4, 8, and 12
Population: The full analysis set included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Parsaclisib
Number analyzed (Participants) | 10
Percentage Change
  Percent change in stimulated salivary flow Week 4: number analyzed (Participants) | 9
  Percent change in stimulated salivary flow Week 4 | 17.57 (36.225)
  Percent change in stimulated salivary flow Week 8: number analyzed (Participants) | 6
  Percent change in stimulated salivary flow Week 8 | -10.59 (32.874)
  Percent change in stimulated salivary flow Week 12: number analyzed (Participants) | 7
  Percent change in stimulated salivary flow Week 12 | -16.07 (41.754)
  Percent change in unstimulated salivary flow Week 4: number analyzed (Participants) | 8
  Percent change in unstimulated salivary flow Week 4 | 228.10 (282.634)
  Percent change in unstimulated salivary flow Week 8: number analyzed (Participants) | 5
  Percent change in unstimulated salivary flow Week 8 | 307.56 (601.557)
  Percent change in unstimulated salivary flow Week 12: number analyzed (Participants) | 6
  Percent change in unstimulated salivary flow Week 12 | 281.12 (541.333)

13. Secondary Outcome: Percentage Change in EULAR Sjögren's Syndrome Disease Activity Index
Description: Defined as percent change in ESSDAI. The ESSDAI is a physician-assessed disease activity index for primary Sjögren's syndrome developed by the EULAR consortium. It consists of 44 items in 12 organ-specific 'domains' contributing to disease activity (constitutional, lymphadenopathy, articular, muscular, cutaneous, glandular, pulmonary, renal, peripheral nervous system, central nervous system, hematological, biological). Each domain is assessed for activity level (i.e., no, low, moderate, high) and assigned a numerical score based on pre-determined weighting of each individual domain. An overall score is then calculated as the sum of all individual weighted domain scores. Overall score is calculated as sum of all individual weighted domain scores (ranges from 0 (best) to 123 (worst activity).
Time Frame: Week 12
Population: Full analysis set included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Parsaclisib
Number analyzed (Participants) | 10
Percentage Change
  Percent Change at Week 4: number analyzed (Participants) | 9
  Percent Change at Week 4 | 1.8 (28.13)
  Percent Change at Week 8: number analyzed (Participants) | 7
  Percent Change at Week 8 | -5.2 (24.09)
  Percent Change at Week 12: number analyzed (Participants) | 7
  Percent Change at Week 12 | -32.1 (25.70)

14. Secondary Outcome: Percentage Change in EULAR Sjögren's Syndrome Patient Reported Index
Description: Defined as percentage change in ESSPRI. EULAR Sjogren's Syndrome Patient-Reported Index (ESSPRI) Score is defined as the change in score between baseline (Week -1) and Week 12. The ESSPRI is a patient-reported, subjective symptom index for primary Sjögren's syndrome developed by the EULAR consortium. It consists of three questions covering the cardinal symptoms of Sjögren's syndrome: dryness, fatigue and pain (articular and/or muscular). Each domain scored on scale of 0-10 (0 =no symptom at all and 10 = worst symptom imaginable), and an overall score is calculated as the mean of the three individual domains where all domains carry the same weight.
Time Frame: Weeks 4, 8, and 12
Population: Full analysis set included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Parsaclisib
Number analyzed (Participants) | 10
Percentage Change
  Percent Change at Week 4: number analyzed (Participants) | 9
  Percent Change at Week 4 | -24.4 (40.36)
  Percent Change at Week 8: number analyzed (Participants) | 7
  Percent Change at Week 8 | -29.0 (28.27)
  Percent Change at Week 12: number analyzed (Participants) | 7
  Percent Change at Week 12 | -25.8 (30.52)

15. Secondary Outcome: Percentage Change in Symptom Scores for Dryness
Description: Defined as percent change in symptom scores for dryness of eyes, mouth, and vagina. The dryness questionnaire will ask participants to rate the dryness of eyes, mouth, or vagina (female participants only) with 24-hour recall using an 11-point numerical rating system ranging from 0 (no dryness) to 10
Time Frame: Weeks 4, 8, and 12.
Population: Full analysis set included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Parsaclisib
Number analyzed (Participants) | 10
Percentage Change
  Percent change in Symptom Score for eye dryness at Week 4: number analyzed (Participants) | 8
  Percent change in Symptom Score for eye dryness at Week 4 | -33.2 (35.29)
  Percent change in Symptom Score for eye dryness at Week 8: number analyzed (Participants) | 6
  Percent change in Symptom Score for eye dryness at Week 8 | -39.3 (23.89)
  Percent change in Symptom Score for eye dryness at Week 12: number analyzed (Participants) | 6
  Percent change in Symptom Score for eye dryness at Week 12 | -40.9 (39.09)
  Percent change in Symptom Score for mouth dryness at Week 4: number analyzed (Participants) | 9
  Percent change in Symptom Score for mouth dryness at Week 4 | -37.7 (37.56)
  Percent change in Symptom Score for mouth dryness at Week 8: number analyzed (Participants) | 7
  Percent change in Symptom Score for mouth dryness at Week 8 | -28.0 (32.97)
  Percent change in Symptom Score for mouth dryness at Week 12: number analyzed (Participants) | 7
  Percent change in Symptom Score for mouth dryness at Week 12 | -50.9 (45.88)
  Percent change in Symptom Score for vaginal dryness at Week 4 | -24.0 (49.18)
  Percent change in Symptom Score for vaginal dryness at Week 8 | -54.2 (51.59)
  Percent change in Symptom Score for vaginal dryness at Week 12 | -49.0 (42.54)

16. Secondary Outcome: Percentage Change in PROMIS Fatigue Short Form
Description: Defined as percent change in PROMIS Fatigue short form. The PROMIS fatigue short form includes 7 items with a rating scale of 1 to 5, 1 being no fatigue and 5 being severe fatigue. The recall period is 7 days.
Time Frame: Weeks 4, 8, and 12
Population: Full analysis set included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Parsaclisib
Number analyzed (Participants) | 10
Percentage Change
  Percent change in Score at Week 4: number analyzed (Participants) | 9
  Percent change in Score at Week 4 | -11.1 (21.87)
  Percent change in Score at Week 8: number analyzed (Participants) | 7
  Percent change in Score at Week 8 | -7.5 (13.17)
  Percent change in Score at Week 12: number analyzed (Participants) | 7
  Percent change in Score at Week 12 | -6.4 (13.16)

17. Secondary Outcome: Female Participants Only : Percentage Change in Female Sexual Function Index
Description: Defined as percent change in FSFI. The FSFI is a brief, self-report measure of female sexual function (female participants only). The questionnaire contains 19 item sexual functioning questionnaire to rate sexual function between 2.0 and 36.0, where 2.0 is low sexual function and 36.0 is high sexual function. Difference in FSFI scores are reported.
Time Frame: Weeks 4, 8, and 12
Population: Full analysis set included all female participants enrolled in the study who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Parsaclisib
Number analyzed (Participants) | 9
Percentage Change
  Percent change in Functional Index at Week 4: number analyzed (Participants) | 8
  Percent change in Functional Index at Week 4 | 39.0 (94.61)
  Percent change in Functional Index at Week 8: number analyzed (Participants) | 6
  Percent change in Functional Index at Week 8 | 8.7 (31.63)
  Percent change in Functional Index at Week 12: number analyzed (Participants) | 6
  Percent change in Functional Index at Week 12 | 23.3 (30.08)

18. Secondary Outcome: Percentage Change in European Quality of Life 5 Dimensions Questionnaire
Description: Defined as percent change in EQ-5D. The EQ-5D is a standardized measure of health status. It consists of 5 questions, each with a 5-item rating scale plus a visual analog scale rating from 1 to 100 for overall health status. Higher score represents more severe symptoms.
Time Frame: Weeks 4, 8, and 12
Population: Full analysis set included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Parsaclisib
Number analyzed (Participants) | 10
Percentage Change
  Percent Change in EQ5D at week 4 | 21.1 (55.37)
  Percent Change in EQ5D at week 8: number analyzed (Participants) | 7
  Percent Change in EQ5D at week 8 | 11.9 (62.91)
  Percent Change in EQ5D at week 12: number analyzed (Participants) | 7
  Percent Change in EQ5D at week 12 | -8.9 (49.54)

ADVERSE EVENTS:
Time Frame: Up to 21 weeks
Arm/Group | Parsaclisib
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 4/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parsaclisib (N=10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT03627065/Prot_001.pdf
  • Statistical Analysis Plan (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/65/NCT03627065/SAP_000.pdf